CLINICAL TRIAL: NCT03395509
Title: Intersectional Screening Program for Diabetes and Cardiovascular Diseases Among 67-years Old Citizens of the Municipal of Viborg
Brief Title: The Intersectional Viborg Screening Program: Cost-(Effectiveness) of Screening for Diabetes and Cardiovascular Diseases
Acronym: VISP
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Annette Langager Hoegh, MD, PhD, Associated professor, Central Jutland Regional Hospital
Other Study IDs: VISP-dk
Record Dates: First submitted 2017-03-15; First posted 2018-01-10 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Aging; Aortic Aneurysm, Abdominal; Hypertension; Mass Screening; Peripheral Arterial Disease; Arrythmia; Diabetes; Carotid Atherosclerosis
Keywords: Mass screening; cardiovascular disease; diabetes
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Hypertension; Peripheral Arterial Disease; Arrhythmias, Cardiac; Diabetes Mellitus; Carotid Artery Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an intersectional and interdisciplinary screening program in Viborg Municipality, including 67 years old citizens. This observational study will estimate the cost-effectiveness of a combined screening program for the following conditions: Abdominal aortic aneurysm, peripheral arterial disease, carotid plaque, hypertension, arrhythmia, and type-2-diabetes. Furthermore, the incidence of the outlined conditions will be described and so will the result of the intervention initiated (secondary medical prophylaxis, smoking cessation, introduction to nutritionally deficient diet etc.)

DETAILED DESCRIPTION:
Description of the cohort: All Viborg municipality citizen are invited to the combined screening program around there 67th birthday. Participants with positive screening results are offered following up consultations and prophylactic interventions are initiated (secondary medical prophylaxis, smoking cessation, introduction to nutritionally deficient diet etc.)

67 years-old citizens from the surrounding municipalities without the offer of the combined screening are used as a control group (1 case: 5 controls).

There are no exclusion criteria.

The screening examination includes: Blood pressure in both arms, ankle brachial blood pressure index (ABI), ultrasound for carotid plaque and abdominal aortic aneurysm, HbA1c and pulmonary function test. Furthermore, a questionnaire on lifestyle parameters, BMI, medical history, walking-related pain and self-rated quality of life (EQ-5D).

One year after the screening examination, the participants will receive a questionnaire in order to evaluate the effect from a participant perspective. The cost(-effectiveness) of the screening program will be estimated after 5 years based on prevalence of diseases, response rate, data extraction from nationwide registries and existing evidence of disease prevention.

ELIGIBILITY:
Inclusion Criteria:

All Viborg municipality citizen are invited to the combined screening program around there 67th birthday.

Exclusion Criteria:

There are no exclusion criteria.

Ages: 67 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All Viborg municipality citizen are invited to the combined screening program around there 67th birthday. Participants with positive screening results are offered following up consultations and prophylactic interventions are initiated (secondary medical prophylaxis, smoking cessation, introduction to nutritionally deficient diet etc.)
  67 years-old citizens from the surrounding municipalities without the offer of the combined screening are used as a control group (1 case: 5 controls).
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Baseline prevalence of peripheral arterial disease (PAD) in men and women aged 67 years from a population screening study on the Municipal of Viborg. | Inclusion will take place from sep. 2014 to sep. 2020
  Ankel Brachial Index
Baseline prevalence of abdominal aortic aneurysm (AAA) | Inclusion will take place from sep. 2014 to sep. 2020
  Ultra sound examination (AP diameter (mm))
Baseline prevalence of diabetes | Inclusion will take place from sep. 2014 to sep. 2020
  Bedside HbA1c
Baseline prevalence of hypertension | Inclusion will take place from sep. 2014 to sep. 2020
  BP(mmhg)
Baseline prevalence of cardiac arrythmia | Inclusion will take place from sep. 2014 to sep. 2020
  ECG
Baseline prevalence of carotic plaques | Inclusion will take place from sep. 2014 to sep. 2020
  Ultra sound examination of A. carotis (IMT in mm)

SECONDARY OUTCOMES:
The cost(-effectiveness) of the screening program | 5 years after ending inclusion
  Socio-economic evaluation (national register data), QALY

CONTACTS AND LOCATIONS:
Overall Officials: Annette Høgh, MD, PhD, Study Chair — Steering Committee; Marie Dahl, MSc(nurse), Study Director — Steering Committee
Locations (1):
- Cardiovascular research Center (KVC), Viborg Hospital, Viborg, Denmark

REFERENCES:
- [Derived] Van Der Giessen D, Hogh A, Svenstrup D, Lindholt JS, Dahl M. Clinical relevance of screening for ECG abnormalities in 67-year-old Danes: a population-based cohort study from the Viborg Screening Programme (VISP). BMJ Open. 2025 Dec 23;15(12):e104169. doi: 10.1136/bmjopen-2025-104169. PMID 41436274
- [Derived] Gras Hojgaard H, Hogh AL, Lindholt JS, Frederiksen K, Dahl M. Effect of nurse-led telephone follow-up to optimize adherence to preventive medication after screen-detected cardiovascular disease: a randomized controlled trial. Eur J Cardiovasc Nurs. 2025 Jul 21;24(5):748-759. doi: 10.1093/eurjcn/zvaf047. PMID 40130283
- [Derived] Andersen JW, Hogh A, Lindholt JS, Sogaard R, Stovring H, Yderstraede KB, Sandbaek A, Dahl M. Impact of Population-Based Screening for Diabetes and Prediabetes Among 67-Year-Olds Using Point-of-Care HbA1c on Healthcare Ultilisation, Results from the VISP Cohort. Clin Epidemiol. 2025 Feb 5;17:75-85. doi: 10.2147/CLEP.S487825. eCollection 2025. PMID 39926308
- [Derived] Dahl M, Andersen JW, Lindholt J, Krarup NT, Borregaard B, Uberg N, Hogh A. Prevalence of interarm blood pressure difference is notably higher in women; the Viborg population-based screening program (VISP). BMC Public Health. 2024 Jul 12;24(1):1868. doi: 10.1186/s12889-024-19388-8. PMID 38997668
- [Derived] Hogh A, Lindholt JS, Sogaard R, Refsgaard J, Svenstrup D, Moeslund NJ, Bredsgaard M, Dahl M. Protocol for a cohort study to evaluate the effectiveness and cost-effectiveness of general population screening for cardiovascular disease: the Viborg Screening Programme (VISP). BMJ Open. 2023 Feb 28;13(2):e063335. doi: 10.1136/bmjopen-2022-063335. PMID 36854592